CLINICAL TRIAL: NCT05674708
Title: Impact of Fat Quality on Postprandial Inflammation (PI:Fat): a Randomized Controlled Trial
Brief Title: Fat Quality and Postprandial Inflammation
Acronym: PI:fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: University of Oslo (Other); Chalmers University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-05898-01
Record Dates: First submitted 2023-01-03; First posted 2023-01-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Response; Inflammation
Keywords: inflammation; diet; fat
MeSH Terms: conditions — Inflammation; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Butter (Active Comparator): Butter based meal
  Interventions: Other: Fat intake
- Coconut (Active Comparator): Coconut based meal
  Interventions: Other: Fat intake
- Corn oil (Active Comparator): Corn oil based meal
  Interventions: Other: Fat intake
- Flax seed oil (Active Comparator): Flax seed oil based meal
  Interventions: Other: Fat intake

INTERVENTIONS:
Other: Fat intake — Four different sources of dietary fat

SUMMARY:
This aim of this randomized controlled postprandial study is to compare the effects of four different far sources (butter, coconut, corn oil and flax seed oil) on postprandial inflammation and metabolic response.

The main questions it aims to answer are:

1. What is the impact of different dietary sources of saturated and polyunsaturated fatty acids on postprandial inflammation?
2. Is the impact of different dietary sources of saturated and polyunsaturated fatty acids on postprandial inflammation mediated by glucose or blood lipids?
3. Can postprandial inflammatory or metabolic response be predicted by individual factors at baseline?

Participants will consume four meals, identical except for the fat source, in random order and sampled for blood and urine for up to 6 hours.

DETAILED DESCRIPTION:
A randomized crossover single meal study will be conducted, comparing four isocaloric meals. The study will be carried out at two sites; one study center is located in Gothenburg, Sweden (Department of Internal Medicine and Clinical Nutrition at the University of Gothenburg) and one study center in Oslo, Norway (Department of Nutrition, University of Oslo).

A total of 20 healthy adults will be recruited and consume four meals, identical except for the fat source, in random order and sampled for blood and urine for up to 6 hours after. Each of the four meals will be separated by a 1 month washout. Subjects will be asked to abstain from rigorous physical activity, alcohol and high-fat foods the day prior to their test meal days.

Four isocaloric high-fat meals with different fatty acid profiles will be compared:

1. butter
2. coconut oil
3. corn oil
4. flax seed oil

At test meal days, study outcomes will be assessed at baseline (0h, fasting, pre meal), 30 min, 1h, 2h, 4h and at 6h (endpoint). At these timepoints, blood pressure will be measured and blood glucose sampled through capillary blood. At baseline, 2h, 4h and 6h, blood will be drawn by venipuncture. Urine will be collected when the participants need to void.

Blood will be collected and handled according to a standardized protocol to prevent any degradation, before stored in -80°C until analysis. At baseline and endpoint, peripheral blood mononuclear cells from blood samples will be isolated using cell preparation tubes and stored at -80 °C until RNA isolation. Lipids, lipoprotein profile and inflammation markers (e.g. cytokines, chemokines, endothelial factors) will be analyzed in samples from 0, 2, 4 and 6 hours.

Differences between meals in the outcomes will be compared using area under the curve and mixed models effect.

ELIGIBILITY:
Inclusion Criteria:

* BMI >18.5
* Willingness to eat study meals

Exclusion Criteria:

* Diabetes
* Cardiovascular disease
* Cancer
* Dyslipidemia
* Anemia (Hb <100)
* Habitual intake of anti-inflammatory drugs
* Recent weight change (>±5%)
* Pregnancy, lactation
* Current smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Inflammation markers | 0, 2, 4 and 6 hours
  Cytokines, chemokines, endothelial factors

SECONDARY OUTCOMES:
Lipoproteins | 0, 2, 4 and 6 hours
  Triglycerides, VLDL
Lipidomics | 0, 2, 4 and 6 hours
  Lipidomics characterization of lipid classes
Blood glucose | 0, 0.5, 1, 2, 4, 6 hours
  Capillary glucose sampling
Blood pressure | 0, 0.5, 1, 2, 4, 6 hours
  Systolic and diastolic
Gene expression | 0 and 4 hours
  Gene expression in peripheral blood mononuclear cells in a subset (N=10) participants

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Bärebring, PhD, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No